CLINICAL TRIAL: NCT01948167
Title: Bending Adolescent Depression Trajectories Through Personalized Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Denver (Other); Rutgers University (Other); University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17-013831; R01MH077178 (NIH)
Record Dates: First submitted 2013-09-18; First posted 2013-09-23 (Estimated); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Depression
Keywords: Depression; Prevention; Adolescents
MeSH Terms: conditions — Depression | interventions — Coping Skills

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interpersonal Psychotherapy- Adolescent Skills Training (Experimental): Interpersonal Psychotherapy- Adolescent Skills Training
  Interventions: Behavioral: Interpersonal Psychotherapy- Adolescent Skills Training
- Coping with Stress (Experimental): Coping with Stress
  Interventions: Behavioral: Coping with Stress

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy- Adolescent Skills Training — A group prevention program that includes a 60-minute pre-group session, 8 weekly 90-minute group sessions, a 60-minute mid-group session, and 3 60-minute booster sessions. IPT-AST focuses on psychoeducation and interpersonal skill-building to decrease interpersonal conflict and increase interpersonal support and competence.
  Other Names: IPT-AST; Teen Talk
  Arms: Interpersonal Psychotherapy- Adolescent Skills Training
Behavioral: Coping with Stress — A group prevention program that consists of 8 acute 90-minute group sessions, 2 parent group sessions, and 3 continuation sessions lasting 60 minutes each. Participants are taught to apply cognitive techniques to their personal thoughts, with the goal of generating effective counterarguments to unrealistic negative beliefs.
  Other Names: CWS
  Arms: Coping with Stress

SUMMARY:
Investigators will combine risk factor research and evidence-based prevention programs, to advance knowledge on personalized approaches to prevention that may be able to better "bend trajectories" of depression that surge throughout adolescence.

DETAILED DESCRIPTION:
Investigators will innovatively combine risk factor research and evidence-based prevention programs, to advance knowledge on personalized approaches to prevention that may be able to better "bend trajectories" of depression that surge throughout adolescence. A randomized controlled trial will examine the benefits of matching youth to two depression prevention programs of Interpersonal Psychotherapy-Adolescent Skills Training (IPT-AST) and Coping with Stress (CWS) for the prevention of depression in adolescents. These two programs are designed to address distinct risk factors for depression - CWS addresses cognitive risks and IPT-AST addresses interpersonal risks. A total of 210 participants across two sites, University of Denver and Rutgers University, will be stratified on cognitive and interpersonal risk and randomized to the two conditions. The goals of the study are to (1) demonstrate that prevention programs can modify depression trajectories among youth by examining within person changes in trajectories over time (three years before and three years after the prevention programs) and by comparing trajectories of prevention youth with changes in same aged cohorts; (2) evaluate a personalized prevention approach to bending depression trajectories by matching and mismatching youth to either CWS or IPT-AST based on individual risk profiles; (3) examine mechanisms of bending depression trajectories and test whether the prevention programs operate via their hypothesized processes; and (4) explore how genetic susceptibility, emotion regulation, and temperament may affect individual response to IPT-AST and CWS. By implementing evidence-based prevention programs after 3-years of prospective naturalistic data collection, this study will contribute essential data on personalized medicine and altering developmental trajectories of first-onset depression.

ELIGIBILITY:
Inclusion Criteria:

* Currently in the 6th to 11th grades
* Adolescent and parent must be English-speaking
* Parental consent and adolescent consent

Exclusion Criteria:

* Presence of current Major Depressive Disorder, dysthymia, bipolar disorder, or significant psychosis
* Suicide attempt in the past week or significant suicidal ideation in the past week
* Presence of significant psychopathology or significant pervasive developmental delays that would make the group inappropriate

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 205 (Actual)
Dates: Start 2013-09; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Presence of a Major Depressive Episode or Dysthymia on the Schedule for Affective Disorders for School Aged Children - Present and Life Time Version (K-SADS-PL) | Post intervention (approximately 3 months post baseline)
  Presence of a depression diagnosis as measured by a semi-structured diagnostic evaluation.
Presence of A Major Depressive Episode or Dysthymia on the Schedule for Affective Disorders for School Aged Children - Present and Life Time Version (K-SADS-PL) | 6-months post-intervention
  Presence of a depression diagnosis as measured by a semi-structured diagnostic evaluation.
Presence of A Major Depressive Episode or Dysthymia on the Schedule for Affective Disorders for School Aged Children - Present and Life Time Version (K-SADS-PL) | 12-months post-intervention
  Presence of a depression diagnosis as measured by a semi-structured diagnostic evaluation.
Presence of A Major Depressive Episode or Dysthymia on the Schedule for Affective Disorders for School Aged Children - Present and Life Time Version (K-SADS-PL) | 18-months post-intervention
  Presence of a depression diagnosis as measured by a semi-structured diagnostic evaluation.
Presence of A Major Depressive Episode or Dysthymia on the Schedule for Affective Disorders for School Aged Children - Present and Life Time Version (K-SADS-PL) | 24-months post-intervention
  Presence of a depression diagnosis as measured by a semi-structured diagnostic evaluation.
Presence of A Major Depressive Episode or Dysthymia on the Schedule for Affective Disorders for School Aged Children - Present and Life Time Version (K-SADS-PL) | 30-months post-intervention
  Presence of a depression diagnosis as measured by a semi-structured diagnostic evaluation.
Presence of A Major Depressive Episode or Dysthymia on the Schedule for Affective Disorders for School Aged Children - Present and Life Time Version (K-SADS-PL) | 36-months post-intervention
  Presence of a depression diagnosis as measured by a semi-structured diagnostic evaluation.
Children's Depression Inventory (CDI) | Post intervention (approximately 3 months after baseline)
  Self-reported depression scores
Children's Depression Inventory (CDI) | 6-months post-intervention
  Self-reported depression scores
Children's Depression Inventory (CDI) | 12-months post-intervention
  Self-reported depression scores
Children's Depression Inventory (CDI) | 18-months post-intervention
  Self-reported depression scores
Children's Depression Inventory (CDI) | 24-months post-intervention
  Self-reported depression scores
Children's Depression Inventory (CDI) | 30-months post-intervention
  Self-reported depression scores
Children's Depression Inventory (CDI) | 36-months post-intervention
  Self-reported depression scores

SECONDARY OUTCOMES:
Children's Global Assessment Scale (CGAS) | Post Intervention (approximately 3 months following baseline)
  Assesses global functioning
Children's Global Assessment Scale (CGAS) | 6-months followup
  Assesses global functioning
Children's Global Assessment Scale (CGAS) | 12-months followup
  Assesses global functioning
Children's Global Assessment Scale (CGAS) | 18-months followup
  Assesses global functioning
Children's Global Assessment Scale (CGAS) | 24-months followup
  Assesses global functioning
Children's Global Assessment Scale (CGAS) | 30-months followup
  Assesses global functioning
Children's Global Assessment Scale (CGAS) | 36-months followup
  Assesses global functioning

CONTACTS AND LOCATIONS:
Overall Officials: Jami F Young, Ph.D., Principal Investigator — Children's Hospital of Philadelphia
Locations (4):
- United States (4):
  - University of Denver, Denver, Colorado
  - University of Illinois Urbana Champaign, Champaign, Illinois
  - Rutgers University, Piscataway, New Jersey
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Jones JD, Schwartz KTG, Davis M, Gallop R, Hankin BL, Young JF. Cognitive and interpersonal moderators of two evidence-based depression prevention programs. J Consult Clin Psychol. 2024 Jul;92(7):432-444. doi: 10.1037/ccp0000886. Epub 2024 Apr 18. PMID 38635190
- [Derived] Young JF, Jones JD, Gallop R, Benas JS, Schueler CM, Garber J, Hankin BL. Personalized Depression Prevention: A Randomized Controlled Trial to Optimize Effects Through Risk-Informed Personalization. J Am Acad Child Adolesc Psychiatry. 2021 Sep;60(9):1116-1126.e1. doi: 10.1016/j.jaac.2020.11.004. Epub 2020 Nov 13. PMID 33189876

DOCUMENTS (1):
  • Informed Consent Form (2017-04-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT01948167/ICF_000.pdf